CLINICAL TRIAL: NCT06261060
Title: Low-Dose Sirolimus to Increase Hematopoietic Function in Patients With RUNX1 Familial Platelet Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0918; NCI-2024-01333 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-02-08; First posted 2024-02-15 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Familial Platelet Disorder; Hematopoietic
MeSH Terms: interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1 (Experimental): Participants will visit the study clinic 2 times during Week 1, one (1) time during Weeks 2-4, and then 1 time every 2 weeks after that (Weeks 6, 8, 10, and so on) until Week 22 (Month 6). Then participants will have a follow-up visit at Week 24 and again at Week 52 (Month 12). Participants will take sirolimus by mouth every day, at about the same time each day. Swallow the tablet(s) whole with a full glass of water (about 1 cup). Do not crush or chew the tablet(s). Participants may take sirolimus with or without food.
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Given by PO

SUMMARY:
To learn about the safety and effects of low-dose sirolimus in participants with RUNX1-FPD.

DETAILED DESCRIPTION:
Primary Objective:

• Evaluate the safety and tolerability of low-dose sirolimus in participants with RUNX1 familial platelet disorder (RUNX1-FPD)

Secondary Objectives:

* Evaluate increases in platelet counts during and after treatment with low-dose sirolimus
* Evaluate changes in somatic mutation variant allele frequency (VAF)
* Monitor the rate of somatic mutation acquisition (ie, mutation burden)
* Assess change in platelet aggregation score
* Measure the change from baseline in bleeding score (ISTH-BAT)
* Evaluate change in mTORC1 downstream signaling (pS6/EBP)

Exploratory Objectives:

* Measure rescue of elevated cytokine profiles
* Evaluate reversal of myeloid skewing using flow cytometry
* Determine changes in bone marrow (eg, megakaryocytic atypia and cellularity)
* Assess changes in patient-reported outcomes measures (eg, EORTC and PRO-CTCAE)
* Describe the pharmacokinetics of sirolimus in patients with RUNX1-FPD
* Determine the correlation between sirolimus trough levels and each endpoint

ELIGIBILITY:
Inclusion Criteria:

* Participants has provided signed, informed consent before initiation of any study specific procedures
* Aged ≥18 years at the time of signing the informed consent
* Confirmed P/LP germline RUNX1 variant per ClinGen Myeloid Malignancy Variant Curation Expert Panel (MM-VCEP) RUNX1-specific variant curation rules80
* Participants must be willing to provide bone marrow sample at time of screening and at the end of treatment with sirolimus
* Platelet count of ≥50,000/µL
* Adequate renal function: estimated glomerular filtration rate based on Modification of Diet in Renal Disease (MDRD) calculation, >30 mL/min/1.73m2
* Adequate hepatic function: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <3 × upper limit of normal (ULN) and total bilirubin <1.5 × ULN
* Adequate cardiac function: left ventricular ejection fraction >50%

Exclusion Criteria:

* Known allergy to sirolimus
* History of lymphoma or other hematologic malignancies
* Uncontrolled bleeding
* Any prior diagnosis of myelodysplastic syndrome or other hematologic malignancy using International Working Group criteria
* Prior treatment with sirolimus or a rapalog, mTOR inhibitor, or B-cell-depleting therapy within 28 days before study day 1
* Treatment with strong inhibitors of cytochrome P450 3A4 (CYP3A4; eg, ketoconazole, voriconazole, itraconazole, erythromycin, telithromycin, and clarithromycin), strong inducers of CYP3A4 (eg, rifampin and rifabutin), other drugs that could increase sirolimus blood concentrations (eg, bromocriptine, cimetidine, cisapride, clotrimazole, danazol, diltiazem, fluconazole, letermovir, protease inhibitors [eg, ritonavir, indinavir, boceprevir, and telaprevir], metoclopramide, nicardipine, troleandomycin, and verapamil), other drugs that could decrease sirolimus blood concentrations (eg, carbamazepine, phenobarbital, phenytoin, rifapentine, St. John's Wort [Hypericum perforatum]), or drugs with blood concentrations that could increase (eg, verapamil) within 7 days before study day 1
* Use of cannabidiol, which can increase blood levels of sirolimus, within 7 days before study day 1
* Myocardial infarction within 6 months before study day 1, congestive heart failure (New York Heart Association > class II)
* Total cholesterol >300 mg/dL or triglyceride >400 mg/dL
* Arterial thrombosis (eg, stroke or transient ischemic attack) within 6 months before study day 1
* Infection requiring intravenous anti-infective treatment within 1 week of study day 1
* Live vaccines (eg, measles, mumps, rubella, oral polio, BCG, yellow fever, varicella, and TY21a typhoid) within 28 days before study day 1
* Known diagnosis of chronic viral infection (eg, hepatitis B or C or HIV, and Epstein-Barr) or tuberculosis
* Women who are pregnant, may become pregnant, or who are breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2026-06-11 (Estimated); Study Completion 2028-06-11 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Courtney DiNardo, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org